CLINICAL TRIAL: NCT00913081
Title: Advancing Niacin by Inhibiting FLUSHing: (ANTI-FLUSH)
Brief Title: Advancing Niacin by Inhibiting Flushing (ANTI-FLUSH)
Acronym: ANTI-FLUSH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB #808911
Record Dates: First submitted 2009-05-29; First posted 2009-06-03 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2011-11

CONDITIONS: Flushing
Keywords: Skin; pharmacology; metabolism; lipid
MeSH Terms: conditions — Flushing | interventions — Quercetin; isoquercitrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Quercetin 500 mg (Experimental): Quercetin 500 mg once, administered one hour before 500 mg immediate-release niacin
  Interventions: Dietary Supplement: Quercetin
- Quercetin 1000 mg (Experimental): Quercetin 1000 mg once, administered one hour before 500 mg immediate-release niacin
  Interventions: Dietary Supplement: Quercetin
- Quercetin 2000 mg (Experimental): Quercetin 2000 mg once, administered one hour before 500 mg immediate-release niacin
  Interventions: Dietary Supplement: Quercetin
- Placebo (Placebo Comparator): Placebo once, administered one hour before 500 mg immediate-release niacin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin — Quercetin 500, 1000, or 2000 mg PO one time
  Other Names: Isoquercetin
  Arms: Quercetin 1000 mg; Quercetin 2000 mg; Quercetin 500 mg
Dietary Supplement: Placebo — Placebo PO one time
  Arms: Placebo

SUMMARY:
Niacin, or vitamin B3, is known to improve cholesterol disorders and is the most effective drug to raise HDL, or the "good cholesterol". The use of niacin has been limited because of a peculiar adverse effect referred to as "flushing', which consists of redness, warmth, tingling and burning. A recent animal study suggests that flavonoids may prevent flushing due to niacin better than drugs like aspirin. The ANTI-FLUSH study is being done to assess whether a presently available dietary supplement known as quercetin, which is a flavonoid, can reduce the flushing that occurs with niacin. We will also assess whether using quercetin to prevent flushing from niacin, can improve how niacin lowers cholesterol.

DETAILED DESCRIPTION:
This study involves people between 21 and 75 years. It will be conducted over a period of 8 weeks, with 4 visits, each separated by 2 weeks. The duration of each visit is 9-10 hours. We will test a different dose of quercetin in each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from the age of 21 to 75, inclusive - 16 subjects, 8 men, 8 women.
2. Ability to understand and agree to informed consent.
3. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

1. Contra-indications or known intolerance to the study medications.
2. History of congestive heart failure, carcinoid, rosacea, renal failure (GFR<60 ml/min/m2).
3. Active liver disease.
4. Active diabetes (defined as any history of type 1 diabetes, or history of type 2 diabetes plus one or more of the following: fasting glucose>= 126mg/dL at screening or use of anti-diabetic medications within 12 months, or glucose>200mg/dL 2 hours after a 75 g oral glucose challenge within 12 months.
5. History of major surgery within the past 6 weeks, or anticipated major surgery during the course of the study, or any history of organ transplant.
6. History of drug abuse within the past 3 years, or regular alcohol use of greater than 14 drinks per week.
7. Women who are pregnant, plan to conceive or lactate.
8. Peri-menopausal women or women currently experiencing flushing.
9. Currently taking vasoactive medications, anti-hypertensives, anti-histamines, Selective Serotonin Re-uptake Inhibitors (SSRIs), NSAIDS, oral steroids, leukotriene inhibitors, supplemental quercetin and > 50mg niacin.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Dunbar, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - CTRC Univ. of Penn - Andrew Mutch Bldg., 4th floor, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled healthy volunteers aged 21 to 75 years. Subjects were recruited at the University of Pennsylvania CTRC following a screening visit to confirm eligibility based on an interview reviewing their health status and medication use, baseline laboratory assessment and the ability to tolerate a 500 mg dose of immediate-release niacin
Pre-assignment Details: Subjects meeting inclusion criteria, able to tolerate 500mg of immediate-release niacin and to provide informed consent were randomized to one of the four study groups. First experimental visit was within 12 weeks of screening visit.
Groups:
- All Study Participants: Participants received one dose of Quercetin 500 mg, Quercetin 100 mg, Quercetin 200 mg, or placebo one hour before immediate-release niacin 500 mg and underwent flushing and pharmacodymic assessments for 8 hours after Quercetin dosing. Each participant then crossed over to one of the remaining dose group/placebo in a randomized, double blind fashion after a washout period of at least 7 days. Each participant received all three doses of Quercetin and placebo.
Period: Quercetin 500 mg + Niacin 500 mg (1day)
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0
Period: Washout #1 (7 Days)
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0
Period: Quercetin 1000 mg + Niacin 500 mg (1day)
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0
Period: Washout #2 (7 Days)
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0
Period: Quercetin 2000 mg + Niacin 500 mg (1day)
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0
Period: Washout #3 (7days)
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0
Period: Placebo + Niacin 500 mg (1day)
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All study participants
Groups:
- All Study Participants: Participants received one dose of Quercetin 500 mg, Quercetin 1000 mg, Quercetin 2000 mg, or placebo one hour before immediate-release niacin 500 mg and underwent flushing and laboratory assessment including plasma free fatty acid, beta-hydroxybutyrate and urinary eicosanoid metabolites for 8 hours after Quercetin dosing. Each participant then crossed over to the next dose group/placebo after a washout period of at least 7 days. Each participant received all three doses of Quercetin and placebo.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Whether Quercetin Dose-dependently Reduces Laser Doppler Flux Index Primary Peak Following Immediate-release Niacin
Description: Laser Doppler flowmetry at the malar eminence measures blood flow quantitatively as red blood cell flux. Flux index is the fold-change in flux over baseline. Flux index primary peak is the maximum flux index between 0-4 hours after niacin.
Time Frame: 8 hour period
Population: All subjects who finished at least one visit were analysed.
Measure: Mean (95% Confidence Interval); unit: Fold change over baseline
Groups:
- Quercetin 500 mg: Participants received one dose of Quercetin 500 mg one hour before immediate-release niacin 500 mg and underwent flushing and laboratory assessment including plasma free fatty acid, beta-hydroxybutyrate and urinary eicosanoid metabolites for 8 hours after Quercetin dosing. Each participant then crossed over to the next dose group/placebo after a washout period of at least 7 days.
- Quercetin 1000 mg: Participants received one dose of Quercetin 1000 mg one hour before immediate-release niacin 500 mg and underwent flushing and laboratory assessment including plasma free fatty acid, beta-hydroxybutyrate and urinary eicosanoid metabolites for 8 hours after Quercetin dosing. Each participant then crossed over to the next dose group/placebo after a washout period of at least 7 days.
- Quercetin 2000 mg: Participants received one dose of Quercetin 2000 mg one hour before immediate-release niacin 500 mg and underwent flushing and laboratory assessment including plasma free fatty acid, beta-hydroxybutyrate and urinary eicosanoid metabolites for 8 hours after Quercetin dosing. Each participant then crossed over to the next dose group/placebo after a washout period of at least 7 days.
- Placebo: Participants received placebo one hour before immediate-release niacin 500 mg and underwent flushing and laboratory assessment including plasma free fatty acid, beta-hydroxybutyrate and urinary eicosanoid metabolites for 8 hours after Quercetin dosing. Each participant then crossed over to the next dose group/placebo after a washout period of at least 7 days.
Arm/Group | Quercetin 500 mg | Quercetin 1000 mg | Quercetin 2000 mg | Placebo
Number analyzed (Participants) | 17 | 17 | 17 | 17
Fold change over baseline | 9.9 [7 to 13] | 9.4 [6 to 12] | 7.7 [5 to 11] | 8.9 [6 to 12]
Statistical Analysis 1: Comparison: Quercetin 500 mg vs Placebo; The null hypothesis is that quercetin, at any dose, does not attenuate niacin-induced increases in dermal blood flow. Because quercetin has not been used to inhibit flushing from niacin in humans, sample size could not be determined statistically. A sample size of 8 men and 8 women was expected to allow separate estimates of effect size, variability, and shape of distribution for men and women; Test type: Superiority or Other; p = 0.5, Mixed Models Analysis
Statistical Analysis 2: Comparison: Quercetin 1000 mg vs Placebo; The null hypothesis is that quercetin, at any dose, does not attenuate niacin-induced increases in dermal blood flow; Test type: Superiority or Other; p = 0.8, Mixed Models Analysis
Statistical Analysis 3: Comparison: Quercetin 2000 mg vs Placebo; The null hypothesis is that quercetin, at any dose, does not attenuate niacin-induced increases in dermal blood flow; Test type: Superiority or Other; p = 0.5, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Quercetin 500 mg | Quercetin 1000 mg | Quercetin 2000 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes